CLINICAL TRIAL: NCT05508061
Title: Fully Automated Glycemic Control With Ultrarapid Insulin in a Bihormonal Closed Loop System in Patients With Type 1 Diabetes
Brief Title: Ultrarapid Insulin Administered by a Bihormonal Closed Loop System in Patients With Type 1 Diabetes
Acronym: FAST 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inreda Diabetic B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL79588.091.22
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
Keywords: Ultra rapid-acting insulin; Lyumjev; Humalog®; Artificial pancreas (AP®); Bihormonal reactive closed loop system; Automated glucose regulation; Time above range
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Allocation by randomization:
  * Study period 1 (Humalog or Lyumjev)
  * Wash-out period (Humalog: standard therapy)
  * Study period 2 (other type of insulin than in Study period 1 (Humalog or Lyumjev))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyumjev (insulin lispro) (Experimental): Administration of Lyumjev for a 30-day study period (dosage and frequency is patient-dependent)
  Interventions: Drug: Insulin Lispro Cartridge [Lyumjev]
- Humalog (insulin lispro) (Active Comparator): Administration of standard used Humalog for a 30-day study period and 8-day wash-out period located between the two study periods (dosage and frequency is patient-dependent)
  Interventions: Drug: Insulin Lispro Cartridge

INTERVENTIONS:
Drug: Insulin Lispro Cartridge [Lyumjev] — Administration of Lyumjev in combination with the AP system
  Other Names: Lyumjev
  Arms: Lyumjev (insulin lispro)
Drug: Insulin Lispro Cartridge — Administration of Humalog in combination with the AP system (standard therapy)
  Other Names: Humalog
  Arms: Humalog (insulin lispro)

SUMMARY:
The main objective is to determine the efficacy of Lyumjev (insulin) in a bi-hormonal reactive closed loop system for automated glucose regulation (artificial pancreas; AP®) in patients with diabetes mellitus type 1. In addition, safety parameters, pharmacodynamics and AP-related parameters will be acquired.

This study is a multicenter, open-label, randomized, cross-over trial in 12 subjects. The subjects will be randomized to receive either Lyumjev or Humalog® for a 30-day study period and will then switch to the alternate insulin treatment after a wash-out period.

DETAILED DESCRIPTION:
Background of the study:

Inreda Diabetic B.V. (Goor, The Netherlands) developed a bi-hormonal reactive closed loop system to automate glucose regulation (artificial pancreas; AP) in patients with diabetes mellitus type 1. In the current CE-marked AP, Humalog® (Eli Lilly) is used as rapid-acting insulin. Currently, the ultra rapid-acting insulin Lyumjev (Eli Lilly) is available but has not yet been tested in combination with the AP of Inreda. Both are insulin lispro, but additions to the insulin lispro allow the insulin to act faster with a shorter duration. The hypothesis is that the combination of Lyumjev and the reactive AP system can decrease the time that glucose values are above range which can have a positive effect on glucose regulation.

Objectives of the study:

The main objective is to determine the efficacy of Lyumjev in the Inreda AP system. Secondary objectives are to assess safety parameters, differences in pharmacodynamics and AP-related outcomes comparing Lyumjev to Humalog®.

Study design:

This study is a multicenter, open-label, randomized, cross-over trial which will be performed in a free-living environment.

Study population:

The study population will comprise 12 subjects with diabetes type 1 using the AP system. Inclusion criteria are subjects from 18 to 75 years and treated with the Inreda AP system for at least 1 month.

Intervention:

The intervention includes the administration of Lyumjev by the Inreda AP system. The subject will be randomized to receive either Lyumjev or Humalog® during the first 30 days. After a wash-out period of 8 days using the standard insulin Humalog®, the subject will switch to the alternate treatment, again for a 30-day period. During the study periods, subjects have to keep a Wi-Fi access point with them.

Primary study parameters/outcome of the study:

Main parameter to express efficacy is the time above range (>10.0 mmol/l), which will be compared between Lyumjev and Humalog®.

Secondary study parameters/outcome of the study:

Safety will be expressed as the side effects of Lyumjev. Pharmacodynamics will be expressed in proportions of time spent in eu-/hypo-/hyperglycemia (%), median glucose value (mmol/l) and glycemic variability (% and interquartile range). These parameters will all be compared between Lyumjev and reference Humalog®.

AP-related outcomes will be expressed in daily administered dosage of insulin and glucagon (units), and the percentage of time that the closed loop algorithm is active (%).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus type 1;
* Treated with the Inreda AP system for a minimum of 1 month;
* Age between 18 and 75 years;
* Willing and able to sign informed consent.

Since subjects are treated with the Inreda AP, the following inclusion criteria will be met:

* Treated with sensor augmented pump (SAP) or CSII for a minimum of 6 months;
* HbA1c < 97 mmol/mol;
* BMI < 35 kg/m^2;
* No use of acetaminophen, as this may influence the sensor glucose measurements.

Exclusion Criteria:

* Impaired awareness of hypoglycemia (score ≥ 4) according to Gold and/or Clarke questionnaire;
* Pregnancy and/or breastfeeding;
* Use of oral antidiabetic agents;
* Insulinoma;
* Hypersensitivity reactions to Lyumjev or any of the excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of time the glucose level is above 10 mmol/l for the study participants | 68 days
  Time the glucose level is above range (>10 mmol/l) expressed as a percentage (%)

SECONDARY OUTCOMES:
Safety parameters | 30 days
  Side effects of Lyumjev
Pharmacodynamic parameters: euglycemia | 68 days
  Percentage of time the glucose level is between 3.9 and 10 mmol/l (%)
Pharmacodynamic parameters: hypoglycemia | 68 days
  Percentage of time the glucose level is below 3.9 mmol/l (%)
Pharmacodynamic parameters: median glucose value | 68 days
  Median of the glucose values (mmol/l)
Pharmacodynamic parameters: standard deviation of glucose value | 68 days
  Standard deviation of the glucose values (parameter required to determine the coefficient of variation)
Pharmacodynamic parameters: mean glucose value | 68 days
  Mean of the glucose values (parameter required to determine the coefficient of variation)
Pharmacodynamic parameters: glycemic variability (CoV) | 68 days
  Glycemic variability expressed as the coefficient of variation (CoV): standard deviation divided by the mean of the glucose values (%)
Pharmacodynamic parameters: glycemic variability (IQR) | 68 days
  Glycemic variability expressed as the interquartile range (IQR) (mmol/l)
AP-related parameters: insulin usage | 68 days
  Daily usage of insulin (units)
AP-related parameters: glucagon usage | 68 days
  Daily usage of glucagon (units)
AP-related parameters: algorithm activity | 68 days
  Percentage of time the algorithm is active (%)

CONTACTS AND LOCATIONS:
Overall Officials: A. van Bon, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Slingeland Hospital, Doetinchem, Gelderland
  - Hospital Gelderse Vallei, Ede, Gelderland

IPD SHARING:
Plan to Share IPD: No